CLINICAL TRIAL: NCT04467190
Title: A Single Visit, Cross-sectional, Observational Study of EBC H2O2 Levels and Other Exhaled Breath Condensate Parameters as Measured by Inflammacheck, in People With a Variety of Respiratory Conditions and Volunteers With no Known Lung Disease
Brief Title: Investigation of Inflammacheck to Measure Exhaled Breath Condensate Hydrogen Peroxide in Respiratory Conditions
Acronym: VICTORY
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/77
Record Dates: First submitted 2020-02-07; First posted 2020-07-10 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People with lung conditions can suffer significantly with their symptoms and often require multiple trips to their GP or secondary care before a diagnosis is made. It can be difficult to diagnose lung disease and to differentiate between different lung conditions, so many people may be misdiagnosed or incorrectly not given a diagnosis. The tests currently used to diagnose lung diseases can be difficult or uncomfortable to do, especially if the person is experiencing lots of symptoms, and therefore can give poor or unreliable results.A new quick and easy to perform test is needed that can differentiate between various lung conditions and people with no lung disease, that can be performed in primary and secondary care with immediate results.

DETAILED DESCRIPTION:
Lung disease is one of the largest contributors to morbidity and mortality in the UK, with 20% of the population diagnosed with, or receiving treatment for a respiratory condition.

Methods of diagnosis are still convoluted and can be difficult to perform, or very costly in patient and clinician time. Some diagnostic tests only look for a specific type of inflammation (e.g. Fractional exhaled Nitric Oxide) and so can overlook other causes. It can be hard to differentiate between different conditions, and as a result there are thousands of people in the UK who have undiagnosed or misdiagnosed respiratory disease.

Measurement of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) is performed during normal tidal breathing, and is well tolerated even in patients with severe airways obstruction and those unable to perform a consistent controlled exhalation. It is also not limited to inflammatory cell specific inflammation.

In studies using the previous version of the Inflammacheck™ device, significant differences have been demonstrated between levels of H2O2 in people with COPD, asthma, ILD and lung cancer compared to healthy controls. These studies have been instrumental in the continued improvement of the device, to ensure that the participant has the best experience, and simplify the procedure, so that the H2O2 result can be obtained with a single test in under 3 minutes.

Although the primary result of the Inflammacheck™ device is EBC H2O2, it is now also able to measure clinically important parameters including breath temperature, humidity, Carbon Dioxide waveforms, and intra-thoracic pressure changes. These parameters, in combination with the EBC H2O2 may be able to be used together to identify differences between people with various respiratory diseases and healthy volunteers. The device has also been improved based on the participant feedback, to ensure that it is user friendly and comfortable.

The investigators need to determine whether the parameters (H2O2, humidity, temperature, exhaled CO2 waveform and intra-thoracic pressure), as measured by 'Inflammacheck™' can either alone or in combination differentiate asthma, COPD, lung cancer, ILD, breathing pattern disorder, bronchiectasis and pneumonia from other each other and from healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged ≥16 years
* A confirmed, clinician made diagnosis of the following (supported by standard accepted diagnostic criteria):
* Asthma with a ≤10 pack year smoking history (confirmed by spirometry and/or airway inflammation and function tests)
* COPD (confirmed by spirometry)
* Bronchiectasis (confirmed by CT scan)
* Interstitial Lung Disease (confirmed by CT scan and MDT/specialist consensus)
* has or is eventually proven to have a histological OR radiological and MDT confirmed diagnosis of primary lung cancer, and not yet started treatment for this
* current pneumonia (confirmed by chest imaging)
* Breathing Pattern Disorder, with no other significant respiratory co-morbidity (specialist confirmed)
* Healthy controls (defined as no current clinical diagnosis of, or be receiving treatment for, a lung or other significant medical disorder).
* Willing and able to give informed consent for participation in the study.
* In a stable state (at least 4 weeks after treatment of an exacerbation of their respiratory disease)

Exclusion Criteria:

* Existing co-morbidities that may prevent them from performing spirometry, for those with asthma, COPD, or healthy controls, with no spirometry in the previous 12 months (at the discretion of the clinical investigator).
* Unable to comprehend the study, provide informed consent, and unable to perform any of the study procedures.
* Requirement of supplemental oxygen (pneumonia participants only)

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants with respiratory disease or healthy controls as defined in the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
To measure the levels of H2O2 in EBC in patients with a range of commonly occurring respiratory conditions | immediately after the procedure (breathing into device)
  levels of H2O2 in Exhaled Breath Condensate
To measure humidity levels in EBC in patients with a range of commonly occurring respiratory conditions | immediately after the procedure (breathing into device)
  level of humidity in breath in Exhaled Breath Condensate
To measure the breath temperature in EBC in patients with a range of commonly occurring respiratory conditions | immediately after the procedure (breathing into device)
  temperature of breath in Exhaled Breath Condensate
To measure CO2 waveform in patients with a range of commonly occurring respiratory conditions | immediately after the procedure (breathing into device)
  exhaled CO2 waveform
To measure intrathoracic pressure in patients with a range of commonly occurring respiratory conditions | immediately after the procedure (breathing into device)
  intrathoracic pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No